CLINICAL TRIAL: NCT01188044
Title: Validating the Use of Accelerometers for the Study of Physical Activity Among Young Malawian Toddlers
Brief Title: Validating Accelerometers to Study Physical Activity of Toddlers
Status: Completed | Type: Observational
Sponsor: Tampere University (Other)
Collaborators: Kamuzu University of Health Sciences (Other); Singapore Clinical Research Institute (Other); University of Glasgow (Other)
Responsible Party: Per Ashorn / Professor of International Health, University of Tampere
Other Study IDs: AG Validation Lungwena
Record Dates: First submitted 2010-08-23; First posted 2010-08-25 (Estimated); Last update posted 2011-01-06 (Estimated); Status verified 2011-01

CONDITIONS: Motor Activity
Keywords: Motor activity; Infant; Validation studies; Malawi; Sub-Saharan Africa
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study group: Healthy children

SUMMARY:
One way to assess impacts of nutrition supplements to health is to measure physical activity. Physical activity can be measured with small devices called "accelerometers". Before they can be used, the devices need to be validated in the population in question. Objectives of this study are to test accelerometers in field conditions and validate their use in 16-18 months old Malawian toddlers. This study does not have a pre-set hypothesis.

DETAILED DESCRIPTION:
Accelerometers have not been validated in children under 2 years of age. In this study 50 toddlers from Lungwena will be recruited. The participants will wear an ActiGraph GT3X+ -accelerometer fitted on their waist with an elastic belt for 7 days. During the measuring, they will have two videotaped one-hour activity observations while wearing and additional accelerometer device fitted on their ankle. The output from the two devices will be compared to observed activity classified with CPAF-method.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent from at least one guardian
* age 16.00 months to 17.99 months
* availability during the period of the study

Exclusion Criteria:

* any guardian reported or observed illness that limits child's physical activity
* a condition reported by the guardian that limits child's activity co-operate in the study
* wasting (weight-for-height < 2 SD)
* concurrent participation in any clinical trial with an intervention

Ages: 16 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy children
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2010-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Feasibility/acceptability | 7-day accelerometer measurement
  Proportion of participants (%) of wearing the accelerometer device for 4 days, 6 hours per day (defined from the accelerometer output data).

SECONDARY OUTCOMES:
Cut-off point values for sedentary, light, moderate, and vigorous activity | First one-hour observation
  Videotaped observation of physical activity is classified by CPAF-method. Vector magnitude of the ActiGraph device attached to hip is compared to this gold standard and cut-off point values are determined by ROC curve analysis. Values are presented in counts/15 seconds. Sensitivity and specificity of the determined cut-point values in predicting the right activity class are also calculated.
Sensitivity and specificity of the determined cut-off point values | Second one-hour observation
  Activity count cut-off points derived from the first one-hour observation are cross-validated by determining their sensitivity and specificity in predicting the right activity class during the second one-hour observation.
Intra- and inter-subject variation in time spent in different activity classes | 7-day accelerometer measurement
  Intra-subject variation in time (%) spent in different activity classes between different days and inter-subject variation in time spent in different activity classes are determined.

CONTACTS AND LOCATIONS:
Overall Officials: Per Ashorn, MD, PhD, Principal Investigator — University of Tampere Medical School; Kenneth Maleta, MBBS, PhD, Principal Investigator — Kamuzu University of Health Sciences; Ashorn Ulla, PhD, Principal Investigator — University of Tampere Medical School
Locations (1):
- University of Malawi, College of Medicine, Mangochi, Malawi

REFERENCES:
- See also: College of Medicine homepage — http://www.medcol.mw/